CLINICAL TRIAL: NCT01051492
Title: Development of Predictive Biomarkers and Novel Approached to Therapy in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: BR07/30/09
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

SUMMARY:
Breast cancer is a common malignancy world-wide, and is the commonest female malignancy in Singapore, with rising trends in incidence over the last 2 decades. While there have been improvements in treatment, mortality from breast cancer remains significant. Development of biomarkers to predict treatment response and toxicity to anti-cancer agents can rationalize the choice of therapy for the individual patients to optimize treatment outcome and to reduce unnecessary toxicities. Development of novel therapies or novel approaches to therapy is also critical to improve the treatment armamentarium in breast cancer. These research strategies will have an significant impact on breast cancer treatment both in Singapore as well as globally.

ELIGIBILITY:
Inclusion Criteria:

This program will recruit mainly cancer patients, predominantly breast cancer patients. The exact inclusion criteria will vary between each individual study. Each individual component study will be submitted to DSRB for separate approval, along with the study protocol and patient informed consent sheet.

Exclusion Criteria:

The exact exclusion criteria will vary between each individual study. Each individual component study will be submitted to DSRB for separate approval, along with the study protocol and patient informed consent sheet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any individual who has been diagnosed with breast cancer
Sampling Method: Non-Probability Sample
Dates: Start 2010-01; Primary Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital Singapore, Singapore, Singapore

REFERENCES:
- [Background] Tan SH, Lee SC, Goh BC, Wong J. Pharmacogenetics in breast cancer therapy. Clin Cancer Res. 2008 Dec 15;14(24):8027-41. doi: 10.1158/1078-0432.CCR-08-0993. PMID 19088019
- [Background] Goetz MP, Rae JM, Suman VJ, Safgren SL, Ames MM, Visscher DW, Reynolds C, Couch FJ, Lingle WL, Flockhart DA, Desta Z, Perez EA, Ingle JN. Pharmacogenetics of tamoxifen biotransformation is associated with clinical outcomes of efficacy and hot flashes. J Clin Oncol. 2005 Dec 20;23(36):9312-8. doi: 10.1200/JCO.2005.03.3266. PMID 16361630